CLINICAL TRIAL: NCT01927016
Title: Factors Linked to Outcomes After Esophageal Cancer Surgery: a Multicenter National Study
Brief Title: Outcomes After Esophageal Cancer Surgery
Acronym: FREGAT I
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: French Eso-Gastric Tumors Working Group (Other); Federation of Research in Surgery (FRENCH) (Other); AFC (Association Francophone de Chirurgie) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2013_01
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Esophageal Neoplasm; Esophageal Disease
Keywords: Esophageal Neoplasm; Esophagus; Surgery; Outcome assessment
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Diseases | interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Esophagectomy for cancer: Patients operated on for a cancer of the esophagus, a Siewert I or II cancer of the oesophago-gastric junction
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Esophagectomy — Esophagectomy for esophageal cancer whatever can be the surgical approach (with or without thoracotomy, minimally invasive or not)

SUMMARY:
Background

* Esophageal carcinoma is the sixth leading cause of cancer -related mortality and the eighth most common cancer worldwide
* The incidence is increasing rapidly
* The overall 5-year survival ranges from 15% to 25% in the literature and poor outcomes are related to diagnosis at advanced stages.
* Surgery used to be the cornerstone of treatment of resectable esophageal cancer, but treatment of esophageal carcinoma remains challenging and need to be considered through a multimodal approach. However the modalities and the impact of this multimodal approach at a national level are unknown Primary objective: To identify predictors of recurrence after esophageal cancer surgery

Secondary objectives :

* 5-year recurrence free survival
* 5-year overall survival
* Predictors of postoperative mortality and morbidity after surgery
* Impact of pCR on recurrence and survival
* Impact of neoadjuvant treatments on recurrence and survival
* Impact of patient preconditioning (such as nutritional support, esophageal prosthesis, mini-invasive approach…) on outcomes

Methodology : European French-speaking retrospective multicentric study Inclusion criteria: All consecutive patients operated on, for a histologically proven carcinoma of the esophagus, the oesophago-gastric junction (Siewert type I and II), in surgical investigator centers between January 2000 and December 2010 Exclusion criteria: Siewert III type carcinoma of the oesophago-gastric junction , non surgical treatment of esophageal carcinoma Planned study period: The data will be collected over a 11-year period from January 2000 to December 2010. Follow up will be ascertained in May 2013.

DETAILED DESCRIPTION:
Patients with an esophageal or junctional carcinoma (including SIewert type I and II) with surgical resection of the primary tumor inclusion date will be date of surgery all patients will be followed during 5 years after surgery or time of death

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients operated on for a cancer of the esophagus , a Siewert I or II cancer of the esopgago-gastric junction in surgical oncology investigator centers
* Surgery performed between 1st January 2000 and 31 December 2010

Exclusion Criteria:

* Siewert III cancer of the oesophago-gastric junction
* Non surgical treatment of the esophageal cancer
* Benign lesion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on for a cancer of the esophagus , a Siewert I or II cancer of the oesophago-gastric junction
Sampling Method: Probability Sample
Enrollment: 2944 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To identify predictors of recurrence after esophageal cancer surgery | 30 May 2012
  clinical factors linked to 5-year recurrence will be identify through univariable and multivariable analysis

SECONDARY OUTCOMES:
5 year recurrence free survival | 30 May 2012
  events: death and recurrence at 5 years after surgery
5 year overall survival | 30 may 2012
  all causes for death at 5 years after surgery
Predictors of postoperative mortality and morbidity after surgery | 30 May 2012
  30-day postoperative mortality and 30-day overall postoperative morbidity
Impact of pCR on recurrence and survival | 30 May 2012
  pathological complete response within the tumor and nodes
Impact of neoadjuvant treatments on recurrence and survival | 30 May 2012
  looking at the impact of neoadjuvant chemo and/or chemoradiation on oncological outcomes
Impact of patient preconditioning (such as nutritional support, esophageal prosthesis, mini-invasive approach…) on outcomes | 30 May 2012
  looking at the impact of nutritional support, endoscopic and surgical procedures on outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Mariette, MD, PhD, Study Director — University Hospital, Lille; Caroline Gronnier, MD, Principal Investigator — CHRU LILLE; Denis Collet, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Bernard Meunier, MD, PhD, Principal Investigator — CHU Rennes
Locations (1):
- University Hospital, Lille, Lille, France

REFERENCES:
- [Derived] Teixeira-Farinha H, Behal H, Cailliau E, Pasquer A, Duhamel A, Thereaux J, Chalret du Rieu M, Lefevre JH, Turner K, Mantziari S, Collet D, Piessen G, Gronnier C; FREGAT Network-AFC Working Group. Impact of primary endoscopic resection on oncological outcomes after esophagectomy for cancer: a retrospective propensity score-based cohort study. Surg Endosc. 2024 Sep;38(9):5169-5177. doi: 10.1007/s00464-024-11077-2. Epub 2024 Jul 22. PMID 39039292
- [Derived] Markar SR, Gronnier C, Duhamel A, Pasquer A, Thereaux J, Chalret du Rieu M, Lefevre JH, Turner K, Luc G, Mariette C; FREGAT Working Group-FRENCH-AFC. Significance of Microscopically Incomplete Resection Margin After Esophagectomy for Esophageal Cancer. Ann Surg. 2016 Apr;263(4):712-8. doi: 10.1097/SLA.0000000000001325. PMID 26135681
- [Derived] Mariette C, Gronnier C, Duhamel A, Mabrut JY, Bail JP, Carrere N, Lefevre JH, Meunier B, Collet D, Piessen G; FREGAT Working Group-FRENCH-AFC; FREGAT Working Group-FRENCH-AFC. Self-expanding covered metallic stent as a bridge to surgery in esophageal cancer: impact on oncologic outcomes. J Am Coll Surg. 2015 Mar;220(3):287-96. doi: 10.1016/j.jamcollsurg.2014.11.028. Epub 2014 Dec 12. PMID 25617915
- [Derived] Gronnier C, Trechot B, Duhamel A, Mabrut JY, Bail JP, Carrere N, Lefevre JH, Brigand C, Vaillant JC, Adham M, Msika S, Demartines N, El Nakadi I, Piessen G, Meunier B, Collet D, Mariette C; FREGAT Working Group-FRENCH-AFC; Luc G, Cabau M, Jougon J, Badic B, Lozach P, Cappeliez S, Lebreton G, Alves A, Flamein R, Pezet D, Pipitone F, Iuga BS, Contival N, Pappalardo E, Mantziari S, Hec F, Vanderbeken M, Tessier W, Briez N, Fredon F, Gainant A, Mathonnet M, Bigourdan JM, Mezoughi S, Ducerf C, Baulieux J, Pasquer A, Baraket O, Poncet G, Vaudoyer D, Enfer J, Villeneuve L, Glehen O, Coste T, Fabre JM, Marchal F, Frisoni R, Ayav A, Brunaud L, Bresler L, Cohen C, Aze O, Venissac N, Pop D, Mouroux J, Donici I, Prudhomme M, Felli E, Lisunfui S, Seman M, Petit GG, Karoui M, Tresallet C, Menegaux F, Hannoun L, Malgras B, Lantuas D, Pautrat K, Pocard M, Valleur P. Impact of neoadjuvant chemoradiotherapy on postoperative outcomes after esophageal cancer resection: results of a European multicenter study. Ann Surg. 2014 Nov;260(5):764-70; discussion 770-1. doi: 10.1097/SLA.0000000000000955. PMID 25379847